CLINICAL TRIAL: NCT05986552
Title: The Influence of Treatment Format on Effectiveness of and Dropout From Schema Therapy for Borderline Personality Disorder: Individual vs. Combined Individual Group Schema Therapy
Brief Title: The Influence of Treatment Format on Schema Therapy for Borderline Personality Disorder
Acronym: IST-IGST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Amsterdam (Other)
Collaborators: Academic Center for Trauma and Personality (Unknown); Arkin Mental Health Care (Unknown)
Responsible Party: Principal Investigator, Arnoud Arntz, Professor, University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMG-4449-2023
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Schema Therapy; Psychotherapy; Therapy format; Randomized Clinical Trial
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Intervention Model Description: Multicenter Randomized Clinical Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessors and investigator are blind to treatment arm up to and including the last follow-up assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Schema Therapy (IST) (Active Comparator): IST will follow the revised protocol described by Arntz & van Genderen. In the first year, 2 sessions (of 50-60 minutes each) per week will be provided, with at least one day in between. In the second year, the frequency will be reduced to once a week for the first 6 months, for the next 3 months to once every two weeks, and for the last 3 months three (booster) sessions will be offered. Therapists need to be trained at least at the junior level of the Dutch ST Association, or of the International ST society (ISST), or having successfully completed the basic IST training and delivering the trial treatments under supervision of a recognized ST supervisor.
  Interventions: Behavioral: Individual Schema Therapy (IST)
- Combined Individual-Group Schema Therapy (IGST) (Active Comparator): In IGST individual sessions (45-60 min) are provided weekly in the first year, and once every 2 weeks in the first three quarters of the second year, after which 3 monthly booster sessions are offered. Group sessions take place once per week for 1.5 years. After 1.5 years, patients leave the group but continue with IST during the last .5 year. If slots are available, new patients can enter the ST group every 10 weeks.
  GST is provided as semi-closed group format developed from the closed format as developed by Farrell & Shaw. IST is based on Arntz & van Genderen, with the addition that IST and GST are coordinated at weekly peer supervision meetings, and that problems related to the patient's participation in the group are put on the IST agenda.
  GST therapists don't need to be IST therapist of their patients. The same training requirements hold as in the IST arm. Additionally, GST-therapists completed GST training and receive(d) at least 10 GST supervisions.
  Interventions: Behavioral: Individual-Group Schema Therapy (IGST)

INTERVENTIONS:
Behavioral: Individual Schema Therapy (IST) — IST is a form of empirically supported specialized psychotherapy for personality disorders. It is delivered in individual sessions by trained therapists.
  Arms: Individual Schema Therapy (IST)
Behavioral: Individual-Group Schema Therapy (IGST) — IGST is a form of empirically supported specialized psychotherapy for personality disorders. It is delivered in the combination of individual sessions and group therapy sessions by trained therapists.
  Arms: Combined Individual-Group Schema Therapy (IGST)

SUMMARY:
The goal of this clinical trial is to compare etc. in patients with borderline personality disorder pure individual schema therapy to combined individual-group schema therapy. The main questions it aims to answer are:

* is there a difference in effectiveness?
* is there a difference in (early) treatment dropout?

Participants will receive either

* individual schema therapy or
* combined individual-group schema therapy.

Researchers will compare individual to combined individual-group schema therapy see if there is a difference in effects and/or a difference in dropout from treatment.

DETAILED DESCRIPTION:
Schema Therapy (ST) for Borderline Personality Disorder (BPD) was originally developed and tested as an individual treatment. Since 2009 group-ST became popular as an supposedly efficient alternative. A RCT found combined individual-group ST to be superior to predominantly group-ST. Thus, individual ST is important. The question arises how combined individual-group ST compares to purely individual ST. This study compares the two formats of ST in a multicenter randomized clinical trial (RCT). The primary outcomes are severity of BPD and (early) treatment dropout. Secondary outcomes include: measures of specific BPD-symptoms; schemas and schema-modes; general mental symptoms; general functioning; and happiness. Moderators hypothesized to predict what patient characteristics are related to differences in effectiveness between the 2 formats are also tested. At least 132 BPD patients from at least 2 sites will be randomized to combined individual-group ST or individual ST. Treatments will take 2 years. Assessments take place every 6 months, and 1 year after end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* BPD as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5), assessed with the Structured Clinical Interview for the DSM-5 Personality Disorders (SCID-5-PD), as primary diagnosis
* BPDSI total score ≥ 20 (i.e, severity in the BPD range, Giesen-Bloo et al., 2010)
* Ability to understand, read, write and speak Dutch, or English if the site has research assistants and therapists of both conditions that are sufficiently fluent in English, as well as an English ST group (as at ACTP).

Exclusion Criteria:

* DSM-5 substance use disorder that needs clinical detox according to the clinical staff (after 6 weeks of abstinence participation is possible).
* Comorbid psychotic disorder (patients with temporary psychotic problems falling under BPD criterion 9 are not excluded)
* DSM-5 Bipolar disorder, type 1 (current or past)
* Acute suicide risk
* Intelligence Quotient (IQ) < 80
* Serious neurological problems such as dementia
* Patients should not start with any form of psychological treatment during screening or during the study's waitlist or treatment. (Low frequency supportive treatment may be continued during wait and screening, but not during the study treatment.)
* Not able or willing to plan participation in the treatment sessions. Note 1. In case of suspicion of exclusion criteria that need specific assessment, like IQ and dementia, a formal diagnostic assessment needs to be done before in/exclusion can be decided.

Note 2. No other psychological treatment during the study follow-up period is provided, unless this is necessary (clinical judgment). The 1 year treatment-free follow-up period is part of the treatment protocol, to help patients gain experience with life without mental health care. After 1 year further treatment can be offered, if indicated.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Borderline Personality Disorder Severity | 0, 6,12,18, 24 and 36 months
  The severity of manifestations of Borderline Personality Disorder during the last 3 months, assessed with a semi-structured clinical interview, the Borderline Personality Disorder Severity Index 5 (BPDSI-5), by an independent trained rater, blind for treatment arm. Minimum score is 0; maximum is 90; higher scores mean worse outcome.
Early treatment dropout rate | 6 months
  Rate of dropout from treatment within the first 6 months

SECONDARY OUTCOMES:
Severity of each of the 9 BPD criteria | 0, 6,12,18, 24 and 36 months
  Severity of separate BPD criteria will be assessed with the subscales of the Borderline Personality Severity Index 5 (BPDSI-5). Each subscale has a range from 0 to 10, higher scores mean worse outcomes.
Suicidality | 0, 6,12,18, 24 and 36 months
  Suicidality will be assessed by the pertinent criterion 5 items of the Borderline Personality Disorder Severity Index 5 (BPDSI-5). The range is 0-10, higher scores mean worse outcomes.
Number of suicide attempts | 0, 6,12,18, 24 and 36 months
  Number of suicide attempts during the last 3 months will be assessed by item 5.13 of the Borderline Personality Disorder Severity Index 5 (BPDSI-5). The minimum is 0, the maximum is not defined. Higher scores mean worse outcomes.
Subjective burden of Borderline Personality Disorder | 0, 6,12,18, 24 and 36 months
  The subjective burden of Borderline Personality Disorder will be assessed with the Borderline Personality Disorder Checklist (BPDCL). The range is 47-235, higher scores mean worse outcome.
General psychopathology symptoms | 0, 6,12,18, 24 and 36 months
  General psychopathology symptoms will be assessed with the Brief Symptom Inventory (BSI). The range is 0-4, higher scores mean worse outcome.
General, social, and societal functioning | 0, 6,12,18, 24 and 36 months
  General, social, and societal functioning will be assessed with the World Health Organization Disability Assessment Schedule (WHODAS), taken by the research assistant who is blind for condition. The minimum score is 0, the maximum 100. Higher scores mean worse outcome.
Happiness | 0, 6,12,18, 24 and 36 months
  Happiness is assessed with the 1-item happiness question validated in more than 30 countries. Range is 1-7, higher scores mean better outcomes.
Early Maladaptive Schemas | 0, 6,12,18, 24 and 36 months
  Early Maladaptive Schemas will be assessed with the Young Schema Questionnaire short form (YSQ-SF). The range is 90-540; higher scores mean worse outcomes.
Schema Modes | 0, 6,12,18, 24 and 36 months
  Schema Modes will be assessed with the Schema Mode Inventory (SMI). The minimum of the dysfunctional mode score is 123, the maximum 738, with higher scores meaning worse outcomes. The minimum of the functional modes score is 20, the maximum 120, with higher scores meaning better outcomes.
Number of medications used | 0, 6,12,18, 24 and 36 months
  Medication use will be monitored during treatment and at each assessment. The minimum number is zero; the maximum is not defined. Higher numbers mean worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Arnoud Arntz, PhD, Principal Investigator — University of Amsterdam; Sophie Rameckers, MSc, Principal Investigator — University of Amsterdam
Locations (2):
- Netherlands (2):
  - Academic Center for Trauma and Personality ACTP, Amsterdam
  - Arkin Mental Health Care, Amsterdam

IPD SHARING:
Plan to Share IPD: No
Given Dutch and European Union legal data protection regulations sharing individual data with other researchers can only be considered if other researchers can guarantee meeting strict conditions.

REFERENCES:
- [Background] Arntz, A. & van Genderen, H. (2020). Schema Therapy for Borderline Personality Disorder, 2nd Edition. Chichester, UK: John Wiley & Sons.
- [Background] Arntz A, Mensink K, Cox WR, Verhoef REJ, van Emmerik AAP, Rameckers SA, Badenbach T, Grasman RPPP. Dropout from psychological treatment for borderline personality disorder: a multilevel survival meta-analysis. Psychol Med. 2023 Feb;53(3):668-686. doi: 10.1017/S0033291722003634. Epub 2022 Dec 1. PMID 36453183
- [Background] Arntz A, Jacob GA, Lee CW, Brand-de Wilde OM, Fassbinder E, Harper RP, Lavender A, Lockwood G, Malogiannis IA, Ruths FA, Schweiger U, Shaw IA, Zarbock G, Farrell JM. Effectiveness of Predominantly Group Schema Therapy and Combined Individual and Group Schema Therapy for Borderline Personality Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Apr 1;79(4):287-299. doi: 10.1001/jamapsychiatry.2022.0010. PMID 35234828
- [Background] Bloo J, Arntz A, Schouten E. The Borderline Personality Disorder Checklist: Psychometric evaluation and factorial structure in clinical and nonclinical samples. Roczniki Psychologiczne // Annals of Psychology. 2017; 20(2): 281-336. http://dx.doi.org/10.18290/rpsych.2017.20.2-3en
- [Background] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612
- [Background] Farrell, J.M. & Shaw, I.A. (2012). Group schema therapy for borderline personality disorder: A step-by-step treatment manual with patient workbook. Hoboken: Wiley.
- [Background] Giesen-Bloo JH, Wachters, LM, Schouten E, Arntz A. The Borderline Personality Disorder Severity Index-IV: Psychometric evaluation and dimensional structure. Personality and Individual Differences. 2010; 49: 136-141.
- [Background] Lobbestael J, van Vreeswijk M, Spinhoven P, Schouten E, Arntz A. Reliability and validity of the short Schema Mode Inventory (SMI). Behav Cogn Psychother. 2010 Jul;38(4):437-58. doi: 10.1017/S1352465810000226. Epub 2010 May 21. PMID 20487590
- [Background] Üstün TB, Kostanjsek, N, Chatterji, S, Rehm, J. Measuring health and disability: manual for WHO disability assessment schedule WHODAS 2.0. Geneva: World Health Organization, 2010.
- [Background] Veenhoven R. World Database of Happiness. 2023. https://worlddatabaseofhappiness.eur.nl/.
- [Background] Young JE, Brown, G. Young Schema Questionnaire-Short Form; Version 3 (YSQ-S3, YSQ) [Database record]. APA PsycTests, 2005. https://doi.org/10.1037/t67023-000